CLINICAL TRIAL: NCT06728137
Title: 2023-05 Rosidal® 1C Pilot Study. Prospective, Mono-centric, Observational Randomized Controlled Study in Healthy Volunteers
Brief Title: Investigation of a New Compression Bandage System Combining Skin Protection, Padding and Compression in One Single Bandage and Comparing to an Existing One-component Bandage.
Status: Recruiting | Type: Observational
Sponsor: Lohmann & Rauscher (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-05
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: prospective; monocentric; randomized controlled trial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers

SUMMARY:
The goal of this study is to learn about the pressure that can be maintained by a new compression bandage over the course of seven days in healthy volunteers. This bandage combines skin protection, padding and compression in one single bandage. It will be applied to the participants lower legs. A similar device will be applied to the other lower leg of the participant. A randomisation method is used for the assignment of the bandages to the participants legs.

Researchers will compare the bandage pressures of both bandages. The so-called sub-bandage pressure will be measured at the day of application and on the next day, the third day and the last day. Participants will also be asked about the wearing comfort of both bandages.

ELIGIBILITY:
Inclusion Criteria:

* Healthy intact skin with no clinical signs of chronic venous insufficiency and no signs of any dermatological condition such as eczema or psoriasis as assessed by investigating physician.
* Ankle circumference > 18 cm (2 cm above ankle) as assessed by the investigating physician.

Exclusion Criteria:

* Known sensitivity to the study products (Rosidal 1C or Urgo K1) or any of their components
* Chronic venous disease with CEAP ≥2
* Ankle Brachial Pressure Index (ABPI) < 0.8 or >1.3
* Ankle circumference <18 or > 32 cm
* Venous echo-Doppler with recognizable abnormalities
* History of

  * malignant ulcer
  * clinically infected wound
  * peripheral arterial occlusive diseases,
  * cardiac insufficiency or cardiac disease such as congestive heart failure, coronary artery disease, myocardial infarction, coronary artery bypass graft
  * cerebrovascular disease
  * liver or renal disease
  * septic phlebitis,
  * phlegmasia coerulea dolens,
  * sensation disorders of the skin
  * eczema, psoriasis
* Use of diuretics, antihypertension or drugs that influence the capillary infiltration
* Comorbidities that could affect compression therapy, particularly diseases causing oedema
* Reliable severe malnutrition
* Diabetes Mellitus
* BMI > 30 kg/m2
* Pregnancy or breast feeding
* Participation in an interventional clinical trial within the last 3 months and during participation in this study
* Participant is analphabet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with static stiffness index SSI ≥ 10 mmHg over the course of 7 days | Day 0, 1, 3, 7
  The pressure is measured underneath the compression bandage ("sub-bandage pressure") which is applied onto the lower leg. A pressure sensor is positioned in between the skin and the compression bandage. The static stiffness index is the pressure difference between active standing and lying.

SECONDARY OUTCOMES:
Percentage of subjects with resting pressures higher than 20 mmHg and 40 mmHg up to day 7 | Day 0, 1, 3, 7
  The resting pressures are obtained during muscle relaxation or rest when the participant is lying.
Rate of participants assessing the wearing comfort on a 6-level scale. | Day 0, 1, 7
  Participants will be asked on their experience on the wearing comfort like mobility of the ankle and slippage or sensations like heat, sweating or pain.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Valentina Dini, Principal Investigator — Department of Clinical and Experimental Medicine, University of Pisa
Locations (1):
- Department of Clinical and Experimental Medicine, University of Pisa, UOC Dermatologia Universitaria, Santa Chiara Hospital AOUP, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dini V, Vietina A, Michelucci A, Rizzello F, Romanelli M, Mosti G, Namislo A, Bohm C, Abel M. A prospective, monocentric, observational randomised controlled pilot study of two all-in-one multicomponent compression systems in healthy volunteers. J Wound Care. 2026 Jan 2;35(1):26-34. doi: 10.12968/jowc.2025.0456. PMID 41528788